CLINICAL TRIAL: NCT05542420
Title: A Multicentre Retrospective Study of Characterization of Treatment Intensified (Add on to Metformin) Real World Adult Population With Type 2 Diabetes Mellitus in India, Pakistan, and Thailand.
Brief Title: A Research Study, Looking at the Characterization of Treatment Intensified (Add on to Metformin) Real-world Adult Population With Type 2 Diabetes Mellitus in India, Pakistan and Thailand.
Acronym: CONVERGE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7528; U1111-1273-4446 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Real world adult population with type 2 diabetes mellitus (T2DM)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — The study will be based on data already recorded in the medical record

SUMMARY:
This study aims to describe demographics, clinical, treatment and healthcare resource utilization characteristics with a particular focus on those relating to cardiovascular disease in selected treatment intensified patients with type 2 diabetes in the real-world settings in India, Pakistan, and Thailand.

The study will be based on data already recorded in participants medical record and no new tests or procedures are required as part of the study.

The study will last for about 6 months and it does not affect participants current treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at type 2 diabetes mellitus (T2DM) diagnosis
3. Year of birth 1928 or later (age blow 90 years old in 2017)
4. T2DM diagnosis in medical record on or after the date of local GLP-1 RA marketing authorization
5. Medical records documenting prior or ongoing treatment with metformin
6. Medical records documenting treatment with other non-metformin T2DM drugs

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
3. Patients with any diagnosis of type 1 diabetes mellitus (T1DM)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with T2DM fulfilling the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
BMI (body mass index) | 6 months prior to Baseline (day 0, defined as the date of first prescription for the most recent antidiabetic medication drug class) (retrospective)
  BMI will be calculated from height and weight data reported as percent of patients
Most recent blood pressure measurement values | 6 months prior to Baseline (day 0, defined as the date of first prescription for the most recent antidiabetic medication drug class) (retrospective)
  Reported as mmHg
The proportion of patients prescribed glucagon-like peptide-1 receptor agonists (GLP-1 RA) | At Baseline (day 0, defined as the date of first prescription for the most recent antidiabetic medication drug class)
  Will be reported as percent of patients
The proportion of patients prescribed cardiovascular disease (CVD) medications | Since the start of medical record
  Will be reported as percent of patients

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Bengaluru, India
- Novo Nordisk Investigational Site, Karachi, Pakistan
- Novo Nordisk Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com